CLINICAL TRIAL: NCT02507388
Title: A Randomized, Double Masked, Three Dose Safety and Pharmacokinetic Study of RTH258 Following Intravitreal (IVT) Injection in Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: Safety and Pharmacokinetics of RTH258 in Subjects With Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RTH258-E003
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-09

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: AMD; nAMD; wetAMD; Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — brolucizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brolucizumab 3 mg (Experimental): Brolucizumab 3 mg/50 μL administered as an intravitreal injection 3 times at 4-week intervals with follow-up for 84 days from the initial injection
  Interventions: Drug: Brolucizumab 3 mg/50 μL
- Brolucizumab 6 mg (Experimental): Brolucizumab 6 mg/50 μL administered as an intravitreal injection 3 times at 4-week intervals with follow-up for 84 days from the initial injection
  Interventions: Drug: Brolucizumab 6 mg/50 μL

INTERVENTIONS:
Drug: Brolucizumab 3 mg/50 μL — Administered as an intravitreal injection
  Other Names: RTH258; ESBA1008
  Arms: Brolucizumab 3 mg
Drug: Brolucizumab 6 mg/50 μL — Administered as an intravitreal injection
  Other Names: RTH258; ESBA1008
  Arms: Brolucizumab 6 mg

SUMMARY:
The purpose of this study is to assess the systemic pharmacokinetics (PK) and safety of 2 different doses of brolucizumab (3 milligrams (mg)/50 microliters (μL) and 6 mg/50 μL) when administered at 4-week intervals for a total of 3 intravitreal injections in subjects with neovascular age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This study has 2 arms with a 1:1 randomization. Randomization will be stratified by Japanese ethnicity. Half of the subjects in each arm will be of Japanese ethnicity. The other half of the subjects in each arm will be non-Japanese. Subjects in both arms will have visits at Screening, Day 0 (Baseline), Day 1 (24 hours post first injection), Day 3, Day 14, Day 21, Day 28, Day 56, Day 57 (24 hours post the injection on Day 56) and Day 84.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent;
* Active choroidal neovascularization (CNV) lesions secondary to AMD that affect the central subfield in the study eye;
* Best Corrected Visual Acuity (BCVA) > 23 letters in the study eye at Baseline;
* 50 years of age or older at the time of Screening.

Exclusion Criteria:

* Any active ocular infection or inflammation;
* Treatment with aflibercept (EYLEA®), bevacizumab (AVASTIN®), ranibizumab (LUCENTIS®), brolucizumab, or an investigational drug for neovascular AMD prior to enrollment in the study, as specified in protocol;
* Ocular surgery in the study eye, as specified in protocol;
* Uncontrolled glaucoma in the study eye, as specified in protocol;
* Use of steroids in the study eye, as specified in protocol;
* Medical conditions that may prevent study completion;
* Pregnant or nursing (lactating) women;
* Women of child-bearing potential unless using contraception;
* Uncontrolled blood pressure, as specified in protocol;
* Other protocol-specified exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2016-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon, A Novartis Division, Study Director — Alcon, A Novartis Division

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 study centers in Japan and 2 study centers in the United States.
Pre-assignment Details: This reporting group includes all subjects who signed an informed consent form and were assigned an identification number (51), minus one subject exited as a screen failure prior to treatment initiation.
Groups:
- Brolucizumab 3 mg: Brolucizumab 3 milligrams (mg)/50 microliters (μL) administered as an intravitreal injection 3 times at 4-week intervals with follow-up for 84 days from the initial injection
Period: Overall Study
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (8.53) | 73.6 (7.09) | 72.4 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 13 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 13 | 25
  Japan | 13 | 12 | 25
Ancestry [Count of Participants; unit: Participants]
  Japanese | 13 | 13 | 26
  Non-Japanese | 12 | 12 | 24
Primary Diagnosis of Neovascular Age-Related Macular Degeneration [Count of Participants; unit: Participants] — As required by the protocol for inclusion in the study
  Participants | 25 | 25 | 50
Pre-dose Anti-Drug Antibody (ADA) Status [Count of Participants; unit: Participants] — A positive ADA titer prior to the first injection is not unexpected, as pre-existing antibodies to biotherapeutic drugs have been detected in drug-naïve subjects for a variety of antibody fragments.
  Participants
    Negative | 11 | 7 | 18
    Positive | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Analyte Serum Concentration [Cmax (ng/mL)]
Description: Serum concentrations at each collection time point were quantitated, where possible, using a validated immunoassay method. These data were analyzed using a noncompartmental pharmacokinetic (PK) method.
Time Frame: Day 0 (predose), 6 hr, 24 hr, 72 hr, 168 hr, 336 hr, 504 hr, 672 hr
Population: The PK analysis set included all subjects who received an intravitreal (IVT) injection with evaluable PK data and with no major protocol deviations that could have had an impact on the PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg
Number analyzed (Participants) | 25 | 25
ng/mL | 20.7 (29.4) | 77.6 (105)

2. Primary Outcome: Time to Reach Maximum Analyte Serum Concentration [Tmax (h)]
Description: as for outcome 1
Time Frame: Day 0 (predose), 6 hr, 24 hr, 72 hr, 168 hr, 336 hr, 504 hr, 672 hr
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg
Number analyzed (Participants) | 25 | 25
hours | 20.3 (24.6) | 17.4 (14.7)

3. Primary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUC0-tlast (ng*h/mL)]
Description: as for outcome 1
Time Frame: Day 0 (predose), 6 hr, 24 hr, 72 hr, 168 hr, 336 hr, 504 hr, 672 hr
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg
Number analyzed (Participants) | 25 | 25
ng*h/mL | 2480 (5470) | 9160 (12300)

4. Primary Outcome: Area Under the Concentration-time Curve From 0 to Infinity [AUC0-inf (ng*h/mL)]
Description: as for outcome 1
Time Frame: Day 0 (predose), 6 hr, 24 hr, 72 hr, 168 hr, 336 hr, 504 hr, 672 hr
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg
Number analyzed (Participants) | 17 | 24
ng*h/mL | 3380 (6860) | 9770 (12600)

5. Primary Outcome: Elimination Half-life in Serum [t1/2 (h)]
Description: as for outcome 1
Time Frame: Day 0 (predose), 6 hr, 24 hr, 72 hr, 168 hr, 336 hr, 504 hr, 672 hr
Population: PK analysis set. Harmonic mean and jackknife estimate of the standard deviation are presented.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg
Number analyzed (Participants) | 18 | 24
hours | 108 (40.7) | 103 (52.5)

6. Primary Outcome: Concentration of RTH258 Obtained 24 Hours Post Day 0 Injection [C24hr (ng/mL)]
Description: Serum concentration at the specified collection time point was quantitated, where possible, using a validated immunoassay method. The data were analyzed using a noncompartmental pharmacokinetic (PK) method.
Time Frame: Day 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg
Number analyzed (Participants) | 24 | 25
ng/mL | 13.5 (20.0) | 65.7 (107)

7. Primary Outcome: Concentration of RTH258 Obtained 24 Hours Post Day 56 Injection [C24hr (ng/mL)]
Description: as for outcome 6
Time Frame: Day 57
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg
Number analyzed (Participants) | 22 | 25
ng/mL | 12.4 (21.8) | 45.0 (59.9)

8. Secondary Outcome: Percentage of Subjects With Positive Anti-drug Antibody (ADA) Status (Test)
Description: A positive ADA status is defined as induced ADA status with ADA negative at predose and with a post-dose titer value increase of 2 or more dilutions at any time point or boosted ADA status with ADA positive at predose and a post-dose titer value increase by more than 3-fold (1 dilution) at any time point.
Time Frame: Day 0 (predose), Day 28, Day 84
Population: PK analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg
Number analyzed (Participants) | 25 | 25
percentage of participants | 16.0 | 4.0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 105 days). AEs are reported as pre-treatment and treatment-emergent.
Description: An adverse event was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. Ocular AEs are presented for both study eye and non-study eye combined.
Groups:
- Pre-Treatment: All subjects who signed an informed consent form and were assigned an identification number (51), minus one subject exited as a screen failure prior to treatment initiation
- Brolucizumab 3 mg: All subjects who received an IVT injection of brolucizumab 3 mg
- Brolucizumab 6 mg: All subjects who received an IVT injection of brolucizumab 6 mg
Arm/Group | Pre-Treatment | Brolucizumab 3 mg | Brolucizumab 6 mg
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/50 | 2/25 | 1/25
Other Adverse Events (participants affected / at risk) | 2/50 | 10/25 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment (N=50) | Brolucizumab 3 mg (N=25) | Brolucizumab 6 mg (N=25)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Endophthalmitis (Eye disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment (N=50) | Brolucizumab 3 mg (N=25) | Brolucizumab 6 mg (N=25)
Conjunctival haemorrhage (Eye disorders) | 0 | 8 | 8
Eye pain (Eye disorders) | 0 | 2 | 1
Foreign body sensation in eyes (Eye disorders) | 0 | 2 | 1
Retinal haemorrhage (Eye disorders) | 2 | 2 | 1
Vitreal cells (Eye disorders) | 0 | 0 | 2
Vitreous floaters (Eye disorders) | 0 | 2 | 4
Nasopharyngitis (Infections and infestations) | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Missing AUCinf and half life values attributable to concentration values below LLOQ may result in biased estimates. Causality assessment of the ADA status is limited due to the high number of subjects with positive ADA at baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.